CLINICAL TRIAL: NCT02701530
Title: Smoking Cessation for Hospital Employees With Low Education in the Capital Region of Denmark. The RESPEKT Study.
Brief Title: Smoking Cessation for Hospital Employees With Low Education.
Acronym: RESPEKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Rygestopkonsulenterne, Hillerød (Unknown); University of Aarhus (Other)
Responsible Party: Principal Investigator, Charlotta Pisinger, Consultant Senior researcher Ass Prof, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F-51061
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted smoking cessation (Experimental): Smoking cessation program tailored in cooperation with the target group; smokers with low education.
  Peer-based anti-relapse strategy. Recruitment strategy: peer-driven, written invitations and posters.
  Interventions: Behavioral: Targeted smoking cessation
- Control (No Intervention): No smoking cessation program.

INTERVENTIONS:
Behavioral: Targeted smoking cessation — Smoking cessation program developed in cooperation with and aimed at smokers with low education.
  Other Names: Smoking cessation - tailored to smokers with low education
  Arms: Targeted smoking cessation

SUMMARY:
The aim of this trial is to develop a new tailored smoking cessation program for smokers with low education. Smokers are involved in design of the intervention. The effect of the intervention is then tested in a randomised controlled trial. Half of workplaces will be offered the intervention and the other half will be control group, not receiving any offer.

DETAILED DESCRIPTION:
The target group of this trial is smokers with low education working in hospitals in the Capital Region of Denmark.

The aim is to develop a new tailored smoking cessation program for and together with smokers with low education. We selected following seven positions/occupations as proxy for low socioeconomic status: cleaner, porter, kitchen staff, social and health care assistant, service assistant, technical staff and medial secretary.

In first step the investigators perform focus group interviews with the target group to identify wishes and barriers. In next step the investigators design the new tailored smoking cessation program together with smokers with low education.

Then the investigators test the effect of the smoking cessation program in a randomised controlled trial. All hospitals in the Capital Region of Denmark except one are included (the last hospital is situated on a remote island). Half of the hospitals are randomised to be intervention group and the other half is control group. Recruitment will be by written invitations, posters and primarily by peer-recruitment (smokers with low education who are ambassadors for the project at the work places). Posters and written invitations show photos of the ambassadors in the target group and their statements; why they have decided to quit smoking.

The group-based smoking cessation intervention is designed with guidance from the anchor persons. There is no moralizing or disease-focusing, few written materials and a lot of drawings and humor. The intervention will be in small groups (4-6 persons), with six sessions (á 1½-2 hours) taking place at the workplace during working time. All counsellors are ex-smokers. Stress-management is included at each session. We offer free nicotine products or varenicline by choice, for up to 12 weeks. Nicotine replacement therapy is always based on the patch and combined with inhaler or mouth spray p.n. Nicotine gum is not offered.

The investigators measure validated abstinence rates at each session and 6 months after last session.

Main end-point is smoking rates after 12 months in intervention hospitals compared with smoking rates in control hospitals.

ELIGIBILITY:
Inclusion Criteria: employee with low education working in an intervention hospital in the Capital Region of Denmark.

We selected following seven positions/occupations as proxy for low socioeconomic status: cleaner, porter, kitchen staff, social and health care assistant, service assistant, technical staff and medial secretary.

-

Exclusion Criteria:

* does not speak Danish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7003 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Smoking rate in hospitals randomised to intervention or control group | 12 months
  Self-reported point abstinence

SECONDARY OUTCOMES:
Smoking cessation rate in persons participating in the group-based intervention | 6 months
  Self-reported point abstinence + carbonmonoxide validated abstinence
Smoking cessation rate in persons participating in the intervention | 6 weeks after fixed quit date
  Carbonmonoxide validated abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Pisinger, MD PhD MPH, Principal Investigator — Research Center for Prevention and Health
Locations (1):
- Research Center for Prevention and Health, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Will be stored in safe database at Research Center for Prevention and Health